CLINICAL TRIAL: NCT06388083
Title: A Phase 1b Open-label Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of Tinlarebant in Japanese Subjects With Stargardt Disease and a Phase 2/3 Randomized, Double-masked, and Placebo-controlled Study to Evaluate the Safety, Tolerability, and Efficacy of Tinlarebant in Subjects With Stargardt Disease
Brief Title: A Phase 2/3 Study to Evaluate the Efficacy and Safety of Tinlarebant in Subjects With Stargardt Disease
Acronym: DRAGON II
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Belite Bio, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LBS-008-CT07
Record Dates: First submitted 2024-04-23; First posted 2024-04-29 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: STGD1; Stargardt Disease 1
MeSH Terms: conditions — Stargardt Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LBS-008, Tinlarebant (Experimental): 5 mg tablet taken orally once a day
  Interventions: Drug: Tinlarebant
- Placebo (Placebo Comparator): Placebo tablets for tinlarebant 5 mg prepared similarly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tinlarebant — 5 mg tablet
  Other Names: LBS-008
  Arms: LBS-008, Tinlarebant
Drug: Placebo — Placebo tablets
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability, and efficacy of tinlarebant in subjects with Stargardt Disease

DETAILED DESCRIPTION:
This study will be comprised of a Phase 1b part conducted in Japan and a Phase 2/3 part. The Phase 1b part of the study will be open-label and will evaluate the pharmacokinetics (PK), pharmacodynamics (PD), safety, and tolerability of daily doses of 5 mg tinlarebant, administered for 7 days, in Japanese subjects with Stargardt Disease (STGD1). The Phase 2/3 part of the study will be randomized, double masked, and placebo controlled to evaluate the safety, tolerability, and efficacy of daily doses of 5 mg tinlarebant, administered for 24 months, in subjects with STGD1.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have clinically diagnosed STGD1 with at least one mutation identified in the ABCA4 gene.
* Subjects must have a defined aggregate atrophic lesion in 1 or both eyes.
* Minimum BCVA is required in the study eye

Exclusion Criteria:

* Any ocular disease other than STGD1 that, in the opinion of the investigator, would complicate assessment of a treatment effect.
* History of ocular surgery in the study eye in the last 3 months.
* Any prior gene therapy.

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
To measure the annualized rate of change from baseline lesion size in aggregate area of atrophy | From baseline to Month 24

SECONDARY OUTCOMES:
To measure the annualized rate of change in total area of atrophy | From baseline to Month 24
Change in BCVA measured by the ETDRS method | From baseline to Month 24

CONTACTS AND LOCATIONS:
Locations (18):
- United States (14):
  - Belite Study Site - US08, Phoenix, Arizona
  - Belite Study Site - US05, La Jolla, California
  - Belite Study Site - US09, San Francisco, California
  - Belite Study Site - US06, Miami, Florida
  - Belite Study Site - US01, Boston, Massachusetts
  - Belite Study Site - US11, Edina, Minnesota
  - Belite Study Site - US04, Rochester, Minnesota
  - Belite Study Site - US14, New York, New York
  - Belite Study Site - US10, Westbury, New York
  - Belite Study Site - US02, Durham, North Carolina
  - Belite Study Site - US07, Philadelphia, Pennsylvania
  - Belite Study Site - US13, Austin, Texas
  - Belite Study Site - US03, Dallas, Texas
  - Belite Study Site - US12, The Woodlands, Texas
- Japan (3):
  - Belite Study Site, Kobe
  - Belite Study Site, Kyoto
  - Belite Study Site, Tokyo
- UK01 Belite Study Site, London, United Kingdom